CLINICAL TRIAL: NCT03629405
Title: Assessment of the Long-Term Efficacy and Barrier Protection of Two Skin Care Products
Brief Title: Assessment of the Efficacy and Barrier Protection of Two Cosmetic Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: proDERM Institut für Angewandte Dermatologische Forschung GmbH (Unknown); Microscopy Services Dähnhardt GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PH4G-04/2016
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Aged Skin
Keywords: pH of the skin; SDS; Lipbarvis; TEWL; Skin hydration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A - Negative control (untreated) for product C (No Intervention): On the forearms four test areas were located, which were labeled from A-D. Test area A contralateral to product C
- B - Negative control (untreated) for product D (No Intervention): On the forearms four test areas were located, which were labeled from A-D. Test area B contralateral to product D
- C - Cosmetic Product WO 3741 with pH 4 (Experimental): On the forearms four test areas were located, which were labeled from A-D. Test area C on the same arm like product D.
  Interventions: Other: C - pH 4 Cosmetic Product WO 3741
- D - Cosmetic Product WO 4081-1 with pH 5.8 (Experimental): On the forearms four test areas were located, which were labeled from A-D.
  Interventions: Other: D - pH 5.8 Cosmetic Product WO 4081-1

INTERVENTIONS:
Other: C - pH 4 Cosmetic Product WO 3741 — Application of the product on the pre-defined skin area on the forearms twice daily for four weeks
  Arms: C - Cosmetic Product WO 3741 with pH 4
Other: D - pH 5.8 Cosmetic Product WO 4081-1 — Application of the product on the pre-defined skin area on the forearms twice daily for four weeks
  Arms: D - Cosmetic Product WO 4081-1 with pH 5.8

SUMMARY:
The aim of the study was to assess the long-term efficacy and barrier protection properties of two cosmetic products on the volar forearms of 20 elderly subjects after four weeks of treatment compared to two untreated test areas.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female and male (at least 30% male subjects)
* From 50 to 75 years of age, equally distributed

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS or infectious hepatitis if known to the subjects
* Conditions which exclude a participation or might influence the test reaction/ evaluation
* Participation or being in the waiting period after participation in similar cosmetic and/or pharmaceutical studies
* Active skin disease at the test area
* One of the following serious illnesses that might require regular systemic medication: insulin-dependent diabetes
* Moles, tattoos, scars, irritated skin, hairs, etc. at the test area that could influence the Investigation

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

PRIMARY OUTCOMES:
Skin pH | baseline, Day 29, Day 30
  Change from baseline at Day 29 and Day 30 of Skin pH Units assessed by pH-meter

SECONDARY OUTCOMES:
Transepidermal Water Loss | baseline, Day 29, Day 30
  Change from baseline at Day 29 and Day 30 of Transepidermal Water Loss (g/m2/h) assessed by Tewameter
Skin Hydration | baseline, Day 29, Day 30
  Change from baseline at Day 29 and Day 30 of Skin Hydration Arbitrary Units assessed by Corneometer
Intercellular lipid lamellae lenght (nm ICLL/1000 nm2 ICS) | baseline, Day 29, Day 30
  Change from baseline at Day 29 and Day 30 of stratum corneum assessed by transmission electron microscopy
Lipid Analysis ((concentration of : Cholesterol (µg/slide), FFA (µg/slide), Ceramide EOS (µg/slide), Ceramide NP (µg/slide), Ceramide NH (µg/slide)) | baseline, Day 29, Day 30
  Change from baseline at Day 29 and Day 30 of corneocyte layer area assessed from the TEM data

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Klaus-Peter Wilhelm, MD, Study Director — proDERM Institute for Applied Dermatological Research, Germany
Locations (1):
- proDERM Institute for Applied Dermatological Research, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No